CLINICAL TRIAL: NCT02540434
Title: Trial of RiaSTAP Versus Cryoprecipitate to Lower Operative Transfusions (TOP-CLOT)
Brief Title: Trial of RiaSTAP Versus Cryoprecipitate to Lower Operative Transfusions
Acronym: TOP-CLOT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility issues prevent completion of recruitment.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1408015402
Record Dates: First submitted 2015-01-28; First posted 2015-09-04 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Coagulopathy
Keywords: Hypofibrinogenemia; ROTEM; Cardiac Surgery; Concentrated Fibrinogen
MeSH Terms: conditions — Hemostatic Disorders; Afibrinogenemia | interventions — cryoprecipitate coagulum; Fibrinogen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- RiaSTAP Arm (Active Comparator): Subjects will be infused with RiaSTAP if the ROTEM FIBTEM A10 value is less than or equal to 10 mm and microvascular bleeding is present.
  Interventions: Device: ROTEM; Drug: RiaSTAP
- Cryopreciptiate Arm (Active Comparator): Subjects will be infused with cryoprecipitate if the ROTEM FIBTEM A10 value is less than or equal to 10 mm and microvascular bleeding is present.
  Interventions: Device: ROTEM; Other: Cryoprecipitate

INTERVENTIONS:
Device: ROTEM — ROTEM delta will be used to identify intraoperative coagulation abnormalities. A blood sample and reagents are placed into a small cup. A pin suspended from a wire is immersed into the sample. The pin rotates back and forth at a fixed angle. The movement of the pin is optically monitored and converted into a real time measurement that is represented graphically. Prior to clot formation, pin rotation is unhindered and is graphically represented as a straight line. As the subject's blood sample starts to clot, strands of clot form between the pin and the cup wall, restricting the movement of the pin depending on the strength of the clot. Graphically, this is represented as a symmetrical widening of the curve.
  Other Names: ROTEM delta
Other: Cryoprecipitate — Subjects with hypofibrinogenemia who are randomized to the Cryoprecipitate arm will be transfused with Cryoprecipitate
  Arms: Cryopreciptiate Arm
Drug: RiaSTAP — Subjects with hypofibrinogenemia who are randomized to the RiaSTAP arm will be transfused with concentrated fibrinogen
  Other Names: Concentrated Fibrinogen
  Arms: RiaSTAP Arm

SUMMARY:
The study aligns with the strategic plan of New York-Presbyterian Hospital (NYPH) to reduce allogeneic blood product use and decrease unnecessary laboratory costs. One of the NYPH Quality and Patient Safety Goals for 2013 was to improve the appropriate use of transfusion guidelines and reduce unnecessary red blood cell (RBC) transfusions. Further, this study will help to answer whether RiaSTAP is a more effective product to treat bleeding than cryoprecipitate. In addition, this trial will provide investigators with preliminary data to apply for future federal funding opportunities, such as the National Heart Lung and Blood Institute sponsored R21 grant (PAR-13-025) that encourages research grant applications from investigators who propose to study research topics in blood banking and transfusion medicine aimed at improving the safety and availability of the blood supply and the practice of transfusion medicine. The investigators anticipate future follow-on studies further investigating fibrinogen concentrate and other similar therapeutics in other perioperative populations, such as in postpartum hemorrhage or surgical ICU settings. Finally, this study involves the use of a safer therapeutic, fibrinogen concentrate, to improve patient care and patient safety. This product does not require the time-intensive process of thawing; therefore, delays in patient care can be avoided by having the product readily available in the OR.

DETAILED DESCRIPTION:
All eligible subjects undergoing cardiac surgery requiring cardiopulmonary bypass (CPB) at New York Presbyterian Hospital-Weill Cornell Medical College will be invited to participate. Consenting subjects will be enrolled and treated according to the protocol. Study investigators anticipate that by consenting all eligible cardiovascular surgical subjects, investigators will not omit the results of subjects who may present with microvascular bleeding after CPB. It is well known that microvascular bleeding occurs more often in reoperations or complex, open cardiac procedures, such as coronary revascularization and valve repair/replacement, or aortic replacements under deep hypothermic circulatory arrest.

Enrolled subjects will receive intraoperative anesthetic, anticoagulation, laboratory testing, and hemodynamic management according to WCMC standards of practice. The need for blood products, including fibrinogen supplementation (CRYO/FIB), will be assessed using a point-of-care (ROTEM) based transfusion algorithm (Appendix A) to ensure consistency and accuracy of treatment. The cardiac anesthesiologists and surgeons are currently using the ROTEM algorithm for the treatment of bleeding during cardiovascular surgery with CPB as part of routine clinical practice at WCMC. The algorithm will have been in place for greater than 9 months prior to study initiation. Randomization will occur in the blood bank when study product (CRYO/FIB) is requested to treat intraoperative acquired hypofibrinogenemia (based on ROTEM tracings). Transfusion of the randomized study product (CRYO/FIB), however, will only occur when the surgeon declares the presence of microvascular bleeding. Surgeons will be blinded to the subject's ROTEM results and randomized study arm. Intraoperative anesthesiologists will not be blinded as the two products require different preparation and administration techniques and cannot be blinded easily.

Once the subject is randomized to their study intervention they will receive that product at all subsequent points during the procedure when fibrinogen replacement is required. If microvascular bleeding occurs and there is no indication by the ROTEM algorithm to administer CRYO/FIB, the subject will revert to standard of care treatment guided by ROTEM or traditional laboratory testing. The subject will not be randomized in the study. In the case of abnormal ROTEM parameters but no clinical evidence of microvascular bleeding as evaluated by the cardiac surgeon, the subject will continue to be monitored carefully for bleeding for the remainder of the procedure. If non-surgical bleeding is subsequently observed prior to chest closure and the consensus is that fibrinogen is needed based on ROTEM results (FIBTEM A10 less than or equal to 10 mm), the subject will be treated with their randomized study product according to the algorithm. Following completion of the procedure, postoperative coagulation management will be according to standard practice and guided by standard laboratory testing, when possible. Unless persistent bleeding is noted, all subjects will receive aspirin (300 mg per rectum) 6 hours postoperatively. Subjects with mechanical or mitral tissue valves will be anticoagulated with warfarin (no heparin bridge) starting on postoperative day two (POD#2). Any subjects experiencing significant arrhythmias (e.g. atrial fibrillation in the perioperative setting) will also be anticoagulated with warfarin. Pharmacologic deep vein thrombosis (DVT) prophylaxis will follow the usual standard of care. Subjects enrolled, randomized, and transfused study product will be observed until hospital discharge (total observation time). Research staff from the Department of Anesthesiology will collect outcomes data, including transfused blood products, laboratory results, evidence of perioperative thrombosis or infection, returns to the OR, length of stay, and mortality using case report forms reports and enter all collected data into a secure REDCap database.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects age 18 and older who have given written informed consent
2. Undergoing cardiac surgery cardiopulmonary bypass (CBP) at Weill Cornell Medical Center

Exclusion Criteria:

1. Subjects on anticoagulation medications including:

   * Clopidogrel, ticagrelor, prasugrel with platelet function analyzer-100 assay closure time (CT) prolonged greater than 15%
   * Last doses of dabigatran, rivaroxaban, apixaban within 72 hours
   * Warfarin with international normalized ratio (INR) greater than 1.5
2. Positive pregnancy test, pregnancy or lactation
3. Thrombocytopenia: platelet count less than 100,000 u/L
4. Emergency procedures
5. Proof or suspicion of a congenital or acquired coagulation disorder (e.g. von Willebrand Factor or via severe liver disease)
6. Participation in another randomized clinical trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos J Skubas, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects undergoing cardiac surgery requiring cardiopulmonary bypass at Weill Cornell Medicine who dont meet exclusion criteria will be invited to participate prior to surgery. They will be recruited after admission to the hospital the day before surgery. If the subject consents to participate, they will be enrolled. Not all will be randomized.
Pre-assignment Details: Enrolled subjects will have initial blood sample taken for baseline ROTEM in the beginning of surgery. During rewarming, the next ROTEM will be run to assess for a FIBTEM A10 < 10. If It is less than/equal to 10, subject will be randomized. If microvascular bleeding is detected subject will get intervention. Note: only 2 subjects were randomized.
Groups:
- Cryopreciptiate Arm: Subjects will be infused with cryoprecipitate if ROTEM FIBTEM A10 value is less than or equal to 10 mm and microvascular bleeding is present.
  ROTEM delta will be used to identify intraoperative coagulation abnormalities. A blood sample and reagents are placed into a small cup. A pin suspended from a wire is immersed into the sample. The pin rotates back and forth at a fixed angle. The movement of the pin is optically monitored and converted into a real time measurement that is represented graphically. Prior to clot formation, pin rotation is unhindered and is graphically represented as a straight line. As the subject's blood sample starts to clot, strands of clot form between the pin and the cup wall, restricting the movement of the pin depending on the strength of the clot. Graphically, this is represented as a symmetrical widening of curve.
  Cryoprecipitate: Subjects with hypofibrinogenemia who are randomized to the Cryoprecipitate arm will be transfused with Cryoprecipitate
Period: Overall Study
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Started (Out of the total 19 subjects that underwent surgery (-3 WD before surgery), only 1 was randomized.) | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: only 1 subject received study intervention (Cryoprecipitate arm). 1 other subject was randomized to receive RiaSTAP, but did not necessitate this intervention so did not get the product. Therefore, the number of participants is marked as 0 for RiaSTAP arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 1 | 1
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Blood Transfusion Total
Description: The combined number of allogeneic blood products (platelets + Fresh Frozen Plasma (FFP) + RBCs) administered to subjects intraoperatively after study intervention.
Time Frame: Procedure length, the average for participants is approximately 6 hours
Population: Only 2 subjects out of total enrolled were randomized. Due to this only 2 subjects being randomized and the study being terminated before completion, no data analysis was done to assess the primary outcome. Therefore there is no measurable data for the mean and SD in either arm.
Groups:
- Cryopreciptiate Arm: Subjects will be infused with cryoprecipitate if the ROTEM FIBTEM A10 value less than or equal to 10 mm and microvascular bleeding is present.
  ROTEM delta will be used to identify intraoperative coagulation abnormalities. A blood sample and reagents are placed into small cup. A pin suspended from a wire is immersed into the sample. The pin rotates back and forth at a fixed angle. The movement of the pin is optically monitored and converted into a real time measurement that is represented graphically. Prior to clot formation, pin rotation is unhindered and is graphically represented as straight line. As the subject's blood sample starts to clot, strands of clot form between the pin and the cup wall, restricting the movement of the pin depending on the strength of the clot. Graphically, this is represented as a symmetrical widening of the curve.
  Cryoprecipitate: Subjects with hypofibrinogenemia who are randomized to the Cryoprecipitate arm will be transfused with Cryoprecipitate
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: 24-hour Blood Transfusion Total
Description: Number of units of RBC, Platelets, cryoprecipitate, FFP, or other blood products administered to subjects receiving study product within the first 24 hours after procedure end
Time Frame: 24 hours
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Groups:
- Cryopreciptiate Arm: Subjects will be infused with cryoprecipitate if the ROTEM FIBTEM A10 value is less than or equal to 10 mm and microvascular bleeding is present. ROTEM delta will be used to identify intraoperative coagulation abnormalities.
  Cryoprecipitate: Subjects with hypofibrinogenemia who are randomized to the Cryoprecipitate arm will be transfused with Cry
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Fibrinogen Repletion
Description: Fibrinogen repletion as measured by ROTEM FIBTEM >10mm after study product administration. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Time Frame: Procedure length, the average for participants is approximately 6 hours
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Incidence of Zero Transfusions
Description: Number of patients who receive no allogeneic blood transfusions following study product administration and first 24 hours after procedure end. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Time Frame: 24 hours
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Correction of Microvascular Bleeding
Description: Difference in surgeon's assessment of microvascular bleeding from approximately 15 minutes before to approximately 15 minutes after administration of study medication. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Time Frame: ~30 min intraoperatively
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: CTICU Length of Stay
Description: Number of days subject spends in cardiothoracic intensive care unit from procedure end to hospital discharge. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Time Frame: Length of Hospital Stay, the average for participants is approximately 7 days
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Hospital Length of Stay
Description: Number of days subject spends in the hospital from procedure end to hospital discharge. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment.
Time Frame: Length of Hospital Stay, the average for participants is approximately 7 days
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Thrombosis and Transfusion Reactions
Description: Incidence of intraoperative or postoperative (during hospital admission only) thrombosis (symptomatic only) and transfusion reactions from procedure to hospital discharge. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment.
Time Frame: Length of Hospital Stay, the average for participants is approximately 7 days
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Infection and Respiratory Failure
Description: Incidence of any infection or respiratory failure from procedure end to hospital discharge. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment.
Time Frame: Length of Hospital Stay, the average for participants is approximately 7 days
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Blood Loss
Description: Quantity of intraoperative and postoperative blood loss as recorded in the anesthesia record and in chest tube outputs (blood drainage volume). Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment.
Time Frame: Length of Hospital Stay, the average for participants is approximately 7 days,
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Incidence of Re-exploration
Description: Incidence of subjects requiring a return to the OR for re-exploration. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment.
Time Frame: Length of Hospital Stay, the average for participants is approximately 7 days
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Mortality Rate
Description: Rate of hospital death during initial hospital admission. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Time Frame: Length of Hospital Stay, the average for participants is approximately 7 days
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Correlation of Laboratory and ROTEM Data
Description: Correlation of fibrinogen, von Willebrand Factor (vWF), and factor VIII levels measured in traditional lab with intraoperative ROTEM parameters. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment.
Time Frame: Procedure length, the average for participants is approximately 6 hours
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Time to Product Administration
Description: Time from request to administration of study product. Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment.
Time Frame: Procedure length, the average for participants is approximately 6 hours
Population: Trial terminated prior to the collection of this data due to feasibility issues preventing completion of recruitment
Arm/Group | RiaSTAP Arm | Cryopreciptiate Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Cryopreciptiate Arm: Subjects will be infused with cryoprecipitate if ROTEM FIBTEM A10 value is less than or equal to 10 mm and microvascular bleeding is present. ROTEM delta will be used to identify intraoperative coagulation abnormalities. Cryoprecipitate: Subjects with hypofibrinogenemia who are randomized to the Cryoprecipitate arm will be transfused with Cryoprecipitate.
  Only enrolled patients randomized to cryoprecipitate arm are at risk for cryoprecipitate-related adverse events. 1 subject out of total 22 consented were randomized to this arm, so 1 subject was at risk to adverse events from this arm. No events were reported.
- RiaSTAP Arm: Subjects will be infused with RiaSTAP if the ROTEM FIBTEM A10 value is less than or equal to 10 mm and microvascular bleeding is present.RiaSTAP: Subjects with hypofibrinogenemia who are randomized to the RiaSTAP arm will be transfused with concentrated fibrinogen.
  Only enrolled patients randomized to RiaSTAP are at risk for riastap-related adverse events. 0 subjects out of total 22 consented were randomized to this arm, so no subjects were at risk to adverse events from this arm.
Arm/Group | Cryopreciptiate Arm | RiaSTAP Arm
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes